CLINICAL TRIAL: NCT07042022
Title: Development of Digital Defocus Vision Training (DDVT) System Based on Virtual Reality Technology and Its Application in Myopia Regulation
Brief Title: Digital Defocus Vision Training (DDVT) System Development and Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, PHD, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023KYPJ282
Record Dates: First submitted 2025-06-07; First posted 2025-06-27 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-06

CONDITIONS: Virtual Reality Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DDVT training group (Experimental): During a six-month follow-up period, participants received 10 minutes of DDVT twice a day (once in the morning, and the other in the afternoon) using a head-mounted virtual reality (VR) display. In daily life during non-training sessions, participants were required to wear frame glasses with complete correction.
  Interventions: Device: Development of digital defocus vision training (DDVT)
- control group (No Intervention): The control group did not have any myopia prevention and control intervention in half a year, and only wore complete-corrected frame glasses in daily life

INTERVENTIONS:
Device: Development of digital defocus vision training (DDVT) — During a six-month follow-up period, participants received 10 minutes of DDVT twice a day (once in the morning, and the other in the afternoon) using a head-mounted VR display. In daily life during non-training sessions, participants were required to wear frame glasses with complete correction.
  Arms: DDVT training group

SUMMARY:
Myopia is the first major disease affecting the visual health of young children. With the increase in the use of electronic products and the decrease in the time for outdoor exercise, the incidence of myopia is increasing year by year. Smith et al. firstly found that peripheral retinal defocus affects the course of myopia development in rhesus monkeys. Subsequent studies have shown that peripheral retinal hyperopic defocus can lead to the growth of the axial length (AL), leading to the development of myopia, while peripheral retinal myopic defocus can effectively slow down the growth of the AL, thus delaying the progression of myopia. Defocus signals can simultaneously change the thickness of the choroid, the vascular tissue behind the retina, and the pigment epithelium, and change the thickness and hardness of the sclera, inhibiting or promoting the growth of the axial length. Therefore, many methods have been designed to intervene in the development of myopia, including orthokeratology and peripheral defocusing glasses. The maintenance process of orthokeratology lens is complex and there is a risk of infection. Peripheral defocus glasses need to be worn for a long time, and the visual quality is unstable. It is still necessary to explore safer, more effective and more practical methods for myopia control. In addition, there may be some correlation between the development of myopia and the decrease of choroidal blood flow. Defocus signal may promote the increase of choroidal blood flow, which may be a way to prevent and control myopia.

Therefore, the investigators integrated the digital defocus paradigm into VR devices and developed a digital defocus vision training (DDVT) system. The purpose of this study was to investigate the effectiveness and safety of DDVT in the prevention and control of myopia in children.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6 to 12 years
* diagnosis of myopia with SER of -0.75 to -6.00 D
* regular astigmatism, and astigmatism less than 2.50D
* anisometropia less than 1.50 D
* a logMAR best-corrected visual acuity (BCVA) of 0.00 or better
* an understanding by participants and their legal guardians of the purpose of the study

Exclusion Criteria:

* other myopia control therapies in the last 6 months (including but not limited to atropine and orthokeratology)
* strabismus, amblyopia, congenital lens dislocation, congenital cataract, glaucoma, uveitis, nystagmus, keratoconus, eye neoplasms and other ocular diseases
* systemic diseases such as nephrotic syndrome or diabetes
* structural changes in the eyeball, a history of ocular surgery or trauma
* other systemic diseases affecting eye health
* participants in other clinical trials at the same time.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
the axial length （AL） | 1 year
  The axial length of the eye is the distance from the anterior surface of the cornea to the posterior surface of the retina. In a normal adult, it is approximately 24 mm , and its growth is closely related to myopia . AL was measured using the IOL Master (Carl Zeiss 500, Meditec, Oberkochen, Germany)

SECONDARY OUTCOMES:
spherical equivalent refraction | 1 year
  Then used 0.5% tropicamide, five minutes apart, to perform three cycloplegia. The pupil is not considered fully dilated until it is larger than 6mm and/or has no light reflex. Autorefraction was measured in each eye using the Topcon KR-8800 (Topcon, Tokyo, Japan). Cycloplegic spherical equivalent refraction (SER) was defined as the spherical degree plus half of the cylindrical degree.

OTHER OUTCOMES:
Negative relative accommodation | 1 year
  Negative relative accommodation (NRA) refers to the degree of relaxation of the eye's accommodation ability when the convergence is fixed. It is one of the important indicators for evaluating binocular visual function. NRA was measured using the Topcon CV-5000 (Topcon, Tokyo, Japan)
Positive relative accommodation | 1 year
  Positive relative accommodation (PRA) refers to the ability of energy regulation to increase when the convergence remains unchanged in the binocular fixation state. It is used to evaluate the accommodative reserve capacity of patients。 PRA was measured using the Topcon CV-5000 (Topcon, Tokyo, Japan)
The accommodation facility | 1 year
  The accommodation facility refers to the ability of the eye to adjust its state quickly as needed, which in the field of vision is expressed as ciliary muscle accommodation speed. The accommodation facility was measured using a ± 2.0 D flipper lens; IOP was measured using the Topcon CT-1 (Topcon, Tokyo, Japan).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Guangdong Provincial Key Laboratory of Ophthalmology and Visual Science, Sun Yat-Sen Universit, Guangzhou, Guangdong
  - Beijing Ophthalmology and Visual Sciences Key Laboratory, Beijing Tongren Eye Center, Beijing